CLINICAL TRIAL: NCT04847648
Title: Air-polishing in the Treatment of Peri-implantitis - a Randomized Controlled Trial
Brief Title: Air-polishing in the Treatment of Peri-implantitis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Principal Investigator, Jan Derks, Associate Professor, Göteborg University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-00169
Record Dates: First submitted 2021-04-07; First posted 2021-04-19 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Peri-Implantitis
Keywords: Non-surgical therapy; Surgical therapy; Air abrasives; Air polishing
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Intervention Model Description: The project will be conducted as a two-armed randomized controlled clinical trial of 5-year duration in three clinical centers.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Clinical assessments will be performed by assessors unaware of group allocation. Bone level changes over time will be assessed on radiographs and expressed in mm by examiners blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - Mechanical instrumentation of implant surface (Active Comparator): The control group will be subjected to non-surgical decontamination including the use of hand instruments and polishing cups aiming at the removal of all supra-mucosal soft and hard deposits from the implant surfaces.
  Interventions: Procedure: Mechanical decontamination
- Test - Mechanical instrumentation and air-polishing of implant surface (Experimental): In the test group the mechanical instrumentation will be supplemented by the use of an air-polishing device during non-surgical therapy.
  Interventions: Procedure: Air-polishing; Procedure: Mechanical decontamination

INTERVENTIONS:
Procedure: Air-polishing — Air-polishing with erythritol powder during non-surgical therapy (at baseline, 5 seconds per surface, and, if necessary, at 3 months).
  Arms: Test - Mechanical instrumentation and air-polishing of implant surface
Procedure: Mechanical decontamination — Mechanical instrumentation of implant surfaces during non-surgical therapy (at baseline and, if necesarry at 3 months) including the use of hand instruments and polishing cups aiming at the removal of all soft and hard deposits from the target implant.

SUMMARY:
The aim of the present study is to evaluate the potential benefit of the adjunctive use of an air-polishing device in the non-surgical treatment of peri-implantitis as compared to mechanical infection control alone. Following establishment of adequate patient-performed infection control, 80 patients diagnosed with moderate/severe peri-implantitis at ≥1 implant will be randomized to one of two groups. Non-surgical will be carried out by experienced operators in three clinical centers and the mechanical instrumentation (control group) will be supplemented by the use of air-polishing with erythritol powder (AirFlow Master, EMS, Nyon, Switzerland) in the test group. The primary outcome assessed is "pocket closure" (ie probing pocket depth ≤5 mm & absence of profuse bleeding on probing) after 6 months. Secondary outcomes include changes of clinical signs of soft tissue inflammation, adverse events and patient-reported outcome measures. Outcomes of non-surgical therapy will be evaluated at 3 and 6 months. Sites with remaining pathology at 6 months will be subjected to surgical therapy. Patients are then provided with personalized maintenance care and followed up to a 5-year evaluation.

DETAILED DESCRIPTION:
The project will be conducted as a two-armed randomized controlled clinical trial of 5-year duration in three clinical centers. 80 systemically healthy patients diagnosed with moderate/severe peri-implantitis at ≥1 implant will be enrolled.

Upon enrolment, all patients will receive instructions in oral hygiene measures until adequate plaque control has been established (Plaque Index ≤20%). If required, supraconstructions will be adjusted to facilitate adequate oral hygiene measures. Thereafter, study participants will be randomized into two groups, stratified for smoking (yes/no) and number of implants in need of treatment (single/multiple).

The control group will be subjected to professionally administered non-surgical, mechanical infection control including the use of hand instruments and polishing cups aiming at the removal of all supra-mucosal soft and hard deposits from the target sites. In the test group the aforementioned treatment will be supplemented by the use of an air-polishing device (AirFlow Master, EMS, Nyon, Switzerland) with a specially designed nozzle for sub-mucosal application (PerioFlow Handpiece, EMS, Nyon, Switzerland). Following local anesthesia, the instrument will be used sub-mucosally at all aspects (ie mesial, distal, buccal, lingual) of the affected implant(s) at a power setting reduced to 60% and with a erythritol powder (14 mikrometer, AirFlow Plus Powder, EMS, Nyon, Switzerland). The handpiece will be guided in a circular motion in a corono-apical direction not in contact with the implant surface. Instrumentation time will be limited to 5 seconds at each aspect. Implant-supported supraconstructions will not be removed for the non-surgical treatment. Patients are recalled two weeks later for assessment of patient-experienced outcomes, professional supramucosal cleaning and reinforcement of oral hygiene.

Peri-implant soft tissues will be evaluated at three months. Implant sites with remaining signs of pathology (PPD ≥6 mm and presence of BOP at ≥3 aspects per implant will be subjected to re-treatment according to the initial allocation. The clinical evaluation will be repeated at 6 months. In case of residual signs of pathology, affected sites will be subjected to surgical therapy of peri-implantitis within the subsequent 4 weeks. Full thickness flaps will be elevated and inflamed tissues will be removed. Mineralized deposits on the implant surfaces will be removed with titanium-coated curettes. Surface decontamination will be performed using a rotating titanium brush under irrigation with saline. No bone recontouring of bony walls is intended. Flaps will be sutured to the level of the bone and sutures will be removed after 2 weeks. Implant-supported supraconstructions will be removed for the surgical intervention, if possible.

Maintenance therapy will be provided at 9 and 12 months and based on individual needs during the subsequent follow-up. A renewed evaluation will be performed at 12 and 18 months. Long-term assessments will be carried out annually from years 3 to 5. Should any implant site present with signs of disease progression (increase of PPD >2 mm and additional bone loss >1 mm compared to baseline) at any of the follow-up examinations, the implant will be exited from the study and appropriate additional therapy will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Probing pocket depth of ≥6 mm
* Bleeding and/or suppuration on probing at ≥3 aspects per implant
* Documented radiographic bone loss of ≥2 mm.

Exclusion Criteria:

* Implants with bone loss ≥80% of implant length will not be considered.
* No medical conditions prohibiting non-surgical/surgical treatment of peri-implantitis
* Implant(s) in function ≥1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-14 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants/implants displaying pocket closure | 3 months
  Pocket closure: Probing pocket depth of ≤5 mm and absence of bleeding on probing at ≥3 aspects per implant and absence of suppuration on probing
Proportion of participants/implants displaying pocket closure | 6 months
  Pocket closure: Probing pocket depth of ≤5 mm and absence of bleeding on probing at ≥3 aspects per implant and absence of suppuration on probing
Proportion of participants/implants displaying pocket closure | 18 months
  Pocket closure: Probing pocket depth of ≤5 mm and absence of bleeding on probing at ≥3 aspects per implant and absence of suppuration on probing
Patient satisfaction assessed by visual analogue scale | 3 months
  Patient satisfaction as assessed on a 100 mm VAS
Patient satisfaction assessed by visual analogue scale | 6 months
  Patient satisfaction as assessed on a 100 mm VAS
Patient satisfaction assessed by visual analogue scale | 18 months
  Patient satisfaction as assessed on a 100 mm VAS

SECONDARY OUTCOMES:
Changes in probing pocket depth | 3 months
  Reductions in PPD relative to baseline
Changes in probing pocket depth | 6 months
  Reductions in PPD relative to baseline
Changes in probing pocket depth | 18 months
  Reductions in PPD relative to baseline
Changes in probing pocket depth | 3 years
  Reductions in PPD relative to baseline
Changes in probing pocket depth | 4 years
  Reductions in PPD relative to baseline
Changes in probing pocket depth | 5 years
  Reductions in PPD relative to baseline
Changes in bleeding on probing | 3 months
  Reductions in BOP relative to baseline
Changes in bleeding on probing | 6 months
  Reductions in BOP relative to baseline
Changes in bleeding on probing | 18 months
  Reductions in BOP relative to baseline
Changes in bleeding on probing | 3 years
  Reductions in BOP relative to baseline
Changes in bleeding on probing | 4 years
  Reductions in BOP relative to baseline
Changes in bleeding on probing | 5 years
  Reductions in BOP relative to baseline
Changes in marginal soft soft tissue levels | 3 months
  Changes in marginal soft soft tissue levels relative to baseline
Changes in marginal soft soft tissue levels | 6 months
  Changes in marginal soft soft tissue levels relative to baseline
Changes in marginal soft soft tissue levels | 18 months
  Changes in marginal soft soft tissue levels relative to baseline
Changes in marginal soft soft tissue levels | 3 years
  Changes in marginal soft soft tissue levels relative to baseline
Changes in marginal soft soft tissue levels | 4 years
  Changes in marginal soft soft tissue levels relative to baseline
Changes in marginal soft soft tissue levels | 5 years
  Changes in marginal soft soft tissue levels relative to baseline
Changes in radiographic bone levels | 6 months
  Changes in radiographic bone levels relative to baseline
Changes in radiographic bone levels | 18 months
  Changes in radiographic bone levels relative to baseline
Changes in radiographic bone levels | 3 years
  Changes in radiographic bone levels relative to baseline
Changes in radiographic bone levels | 5 years
  Changes in radiographic bone levels relative to baseline
Rate of adverse events | 3 months
  Emphysema
Rate of adverse events | 6 months
  Emphysema
Rate of adverse events | 18 months
  Emphysema
Patient discomfort as expressed on a visual analogue scale | 3.5 months
  Patient discomfort 2 weeks after non-surgical treatment as expressed on a 100 mm VAS
Patient discomfort as expressed on a visual analogue scale | 6.5 months
  Patient discomfort 2 weeks after surgical treatment as expressed on a 100 mm VAS
Esthetic appreciation as expressed on a visual analogue scale | 3 months
  Esthetic appreciation as expressed on a 100 mm VAS
Esthetic appreciation as expressed on a visual analogue scale | 6 months
  Esthetic appreciation as expressed on a 100 mm VAS
Esthetic appreciation as expressed on a visual analogue scale | 18 months
  Esthetic appreciation as expressed on a 100 mm VAS

CONTACTS AND LOCATIONS:
Overall Officials: Kostas Bougas, PhD, Study Director — Göteborg University
Locations (1):
- Department of Periodontology, Institute of Odontology, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No